CLINICAL TRIAL: NCT07348614
Title: Flex Appeal: A Prospective Randomized Controlled Trial Evaluating the Efficacy of Anesthetic Techniques for Manipulation of Knees Under Anesthesia (MUA)
Brief Title: Flex Appeal: Evaluating the Efficacy of Anesthetic Techniques for Manipulation of Knees Under Anesthesia
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00118605
Record Dates: First submitted 2026-01-14; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Knee Stiffness After Total Knee Arthroplasty
Keywords: knee arthroplasty; spinal anesthesia; general anesthesia
MeSH Terms: interventions — Anesthesia, Spinal; Anesthesia, General; Propofol; chloroprocaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Investigator and surgeon will be masked
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spinal Anesthesia (Experimental): Patients receive spinal anesthesia during MUA (manipulation under anesthesia).
  Interventions: Procedure: Spinal Anesthesia; Drug: Chloroprocaine
- General Anesthesia (Active Comparator): Patients receive general anesthesia during MUA (manipulation under anesthesia).
  Interventions: Procedure: General Anesthesia; Drug: Propofol

INTERVENTIONS:
Procedure: Spinal Anesthesia — Administration of spinal anesthesia for knee manipulation.
  Arms: Spinal Anesthesia
Procedure: General Anesthesia — Administration of general anesthesia for knee manipulation.
  Arms: General Anesthesia
Drug: Propofol — Patients undergoing general anesthesia will receive an induction dose of propofol that will be titrated to effect, and airway support as needed until the patient is appropriately anesthetized for the procedure as determined by the anesthesia and surgical care teams.
  Arms: General Anesthesia
Drug: Chloroprocaine — Patients undergoing spinal anesthesia will receive a spinal injection under standard aseptic technique, with 45mg chloroprocaine.
  Arms: Spinal Anesthesia

SUMMARY:
The purpose of this study is to determine if changing the type of anesthesia improves the outcomes of manipulation and pain control after the procedure. The study will compare a spinal anesthesia with a general anesthesia, to see if there is a better outcome from either anesthesia type.

ELIGIBILITY:
Inclusion:

1. Patients ≥18 years presenting for a manipulation of knee joint under anesthesia.
2. ASA Classification I - III.
3. English speaking patients.

Exclusion:

1. ASA 4 or 5
2. Daily chronic opioid use (over 3 months of continuous opioid use).
3. Inability to communicate pain scores or need for analgesia.
4. Infection at the site of block placement
5. Age under 18 years old or greater than 75 years old
6. Pregnant women (as determined by point-of-care serum bHCG)
7. Intolerance/allergy to local anesthetics
8. Weight <50 kg
9. Suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
10. Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the investigator, may interfere with study assessments or compliance.
11. Current or historical evidence of any clinically significant disease or condition that, in the opinion of the investigator, may increase the risk of surgery or complicate the subject's postoperative course.
12. BMI >50 kg/m2.
13. Allergy or contraindication to local anesthetics or any component of the multimodal analgesic regimen

    (NSAIDs and acetaminophen)
14. Contraindication to spinal injection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change in degrees of motion of the affected knee | At time of procedure completion

SECONDARY OUTCOMES:
Change in pain | Baseline, 24 hours, 48 hours, 72 hours post-procedure
  Participants will be asked to rate pain on a scale of 0-10 with 0 being no pain and 10 being the worst possible pain.
Opioid use in PACU | Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Emily Hall, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: No